CLINICAL TRIAL: NCT02197936
Title: Norwegian Adenomyosis Study: Pathophysiology, Peristalsis, Expression Profiling and Diagnostics, Part III
Brief Title: Norwegian Adenomyosis Study III: Peristalsis
Acronym: NAPPEDIII
Status: Terminated | Type: Observational
Why Stopped: Study was suspended due to organisational difficulties.
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Departement of Biomedical Engineering, Tel Aviv University, Tel Aviv, Israel (Unknown); Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Tina Tellum, Medical Doctor, Oslo University Hospital
Other Study IDs: 2014/637c
Record Dates: First submitted 2014-07-17; First posted 2014-07-23 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Adenomyosis; Infertility; Dysmenorrhea
Keywords: Peristalsis; ultrasound
MeSH Terms: conditions — Adenomyosis; Infertility; Dysmenorrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Peristalsis adenomyosis: with adenomyosis
- Peristalsis control: No adenomyosis

SUMMARY:
Spontaneous contractions (peristalsis) of the non-pregnant uterus is widely investigated and the role of correct peristalsis is most important for correct sperm transport towards the fallopian tubes and implantation of the embryo, thus obtaining pregnancy. At the same time, an impaired uterine peristalsis is discussed to be the reason for lower pregnancy rates and may also account for heavy menstrual bleedings and menstrual pain.

In this study, the uterine peristalsis of women with adenomyosis will be investigated. This condition is associated to heavy menstrual bleeding, menstrual pain and infertility.

DETAILED DESCRIPTION:
The peristalsis of the non-pregnant uterus is widely investigated and the role of correct peristalsis seems to be most important for correct sperm transport towards the fallopian tubes and implantation of the embryo. At the same time, an impaired uterine peristalsis is discussed to be the reason for lower pregnancy rates and may account for dysmenorrhea and menorrhagia. The connection of impaired peristalsis and various clinical symptoms has been shown for patients with e.g. leiomyoma and endometriosis, but not for women with adenomyosis, though the concept seems to be widely accepted.

It has also been repeatedly postulated that impaired peristalsis interferes with implantation of the embryo, yet Martinez-Conejero published a trial that showed a higher incidence of miscarriage, but no effect on embryo implantation in women undergoing oocyte donation. This might either indicate that the postulated effect of peristalsis is wrong or, more likely, since this is a study in an IVF setting, that hormonal treatment with gonadotropin-releasing hormone (GnRH)-agonist could improve implantation.

It is possible to monitor peristalsis with transvaginal ultrasound and standard patterns of uterine peristalsis are defined by Jiland already in 1996.

Findings resulting from the investigations in this study may help to determine the role and extent of impaired peristalsis in women with adenomyosis and possibly give new clues on potential treatments, as well as fill a gap in today's knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged 20-45 years having been diagnosed with adenomyosis earlier and have no other pathology of the uterus, regardless of clinical symptoms.

Exclusion Criteria:

* Postmenopausal women,
* Pregnant women,
* Gynaecological cancer,
* GnRH analog therapy or systemic hormone therapy in the last three months prior to hysterectomy,
* Endometriosis,
* Uterine fibroids

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women suffering from adenomyosis and healthy control group
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2014-07; Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Frequency of peristaltic waves in Hz | five minutes
  Frequencies of peristalsis in patients with and without adenomyosis will be compared.
Altitude of peristaltic waves in mm | five minutes
  The altitude of the peristaltic waves in patients with and without adenomyosis will so be compared.

SECONDARY OUTCOMES:
direction of uterine peristalsis: antegrade, retrograde | 5 minutes, at time of ovulation
  Dynamic motility characterization of the uterine peristalsis in women with adenomyosis.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Tellum, MD, Principal Investigator — Oslo University Hospital, Ullevål; Marit Lieng, PhD, MD, Study Chair — Oslo University Hospital
Locations (1):
- Department of Gynecology, Oslo University Hospital Ullevål and Rikshospital, Oslo, Norway